CLINICAL TRIAL: NCT06659224
Title: The Risk of Developing Acute Myeloid Leukaemia in Patients With Ewing's Sarcoma: A SEER-based Study
Brief Title: The Risk of Acute Myeloid Leukaemia in Patients With Ewing's Sarcoma
Status: Completed | Type: Observational
Sponsor: asmaa salama ibrahim (Other)
Responsible Party: Sponsor-Investigator, asmaa salama ibrahim, Resident physician of gastroenterology, Suez Canal University
Organization: Suez Canal University (Other)
Other Study IDs: A275
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia (AML); Ewing Sarcoma
Keywords: acute myeloid leukemia; Ewing sarcoma; SEER
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Ewing's sarcoma is an uncommon yet vital malignancy of bone. It demonstrates a predilection for the pediatric and young adult population. Chemotherapy is considered an important treatment modality for Ewing's sarcoma. However, the development of therapy-related leukemia, especially acute myeloid leukemia following treatment, is attributed to the use of substances such as alkylating agents and topoisomerase inhibitors which are genotoxic. There is a very few studies elaborating on the incidence rates of such complications. So, our aim is to quantify the risk of developing acute myeloid leukemia in Ewing sarcoma patients and provide an updated evidence to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Ewing sarcoma
* Latency exclusion period of 6 months
* Sequence 0 or 1

Exclusion Criteria:

* patients lacking age documentation or age reported only on death certificates or autopsies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Ewing sarcoma between 2000 and 2021, followed up for more than 10 years after the initial diagnosis. Site record ICD-O-3/WHO 2008 restricted to bone and soft tissue; and histological type ICD-O-3 specified as Ewing sarcoma (9364)
Sampling Method: Probability Sample
Enrollment: 2631 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The standardized incidence ratio and excess risk of developing acute myeloid leukemia in Ewing's sarcoma patients | from Jan, 2000 till Dec, 2021
  The surveillance, epidemiology and End Results (SEER) database was used to calculate the standardized incidence ratio (SIR) as Observed/Expected (O/E) and calculated the excess absolute risk for acute myeloid leukemia in Ewing's sarcoma patients.

SECONDARY OUTCOMES:
The standardized incidence ratio and excess risk of second primary malignancies in Ewing's sarcoma patients across different racial groups | from Jan, 2000 till Dec, 2021
The standardized incidence ratio and excess risk of second primary malignancies in Ewing's sarcoma patients between different stages | from Jan, 2000 till Dec, 2021

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Ellaithy, MD, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided